CLINICAL TRIAL: NCT06066242
Title: Optimizing Induction Chemotherapy Regimens for Newly Diagnosed Elderly Acute Myeloid Leukemia Patients Who Are Eligible for Intense Chemotherapy: A Multicenter, Randomized, Controlled Phase II Clinical Trial
Brief Title: Optimizing Induction Chemotherapy Regimens for ND Elderly AML Patients Who Are Eligible for Intense Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023059
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: elderly; newly diagnosed; fit; induction regimen
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AZA+VEN (Experimental): Two courses of azacitidine combined with venetoclax as induction regimen
  Interventions: Other: Different induction chemotherapy regimens
- DA/IA 3+7 (Experimental): Daunorubicin or Idarubicin ×3 days combined with cytarabine × 7 days as induction regimen
  Interventions: Other: Different induction chemotherapy regimens
- DA/IA 2+5+VEN (Experimental): Daunorubicin or Idarubicin ×2 days, cytarabine × 5 days combined with venetoclax as induction regimen
  Interventions: Other: Different induction chemotherapy regimens

INTERVENTIONS:
Other: Different induction chemotherapy regimens — azacitidine combined with venetoclax or chemotherapy with or without venetoclax

SUMMARY:
The optimal induction chemotherapy regimen for newly diagnosed elderly AML patients who are eligible for intense chemotherapy is currently not well defined. Thus, we intend to conduct a multicenter, randomized, controlled clinical trial to compare the safety and efficacy of three different induction regimens (Ven+AZA vs DA/IA 3+7 vs DA/IA 2+5+VEN). A total of 90 patients will be enrolled in this study and segregated into thress groups with 30 in each group. Patients who achieve CR/CRi/CRh after using different induction regimens will receive the same consolidation and maintenance therapy. Allogeneic hematopoietic stem cell transplantation is recommended for patients in the high-risk group or those with persist MRD positivity. After completion of the treatment phase, patients entered the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study and voluntarily sign informed consent.
2. Age: 60~75 years old, gender unlimited.
3. Patients diagnosed with acute myeloid leukemia according to "The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia" who haven't been treated.
4. Eastern Cooperative Oncology Group (ECOG) physical state score: 0-2.
5. Fit for intensive chemotherapy.
6. The function of main organs should meet the following standards before treatment: Kidney: serum creatinine ≤ 2× upper limit of normal range (ULN); Liver: total bilirubin ≤ 1.5 × ULN, AST and ALT ≤ 2.5× ULN; Heart: myocardial enzymes ≤ 2× ULN and normal ejection fraction by cardiac color doppler ultrasound

Exclusion Criteria:

1. Patients with acute promyelocytic leukemia
2. Patients with RUNX1::RUNX1T1 or CBFB::MYH11 fusion gene
3. Patients with BCR::ABL fusion gene
4. Patients who have received a prior treatment for AML with chemotherapy, hypomethylating agents or venetoclax before.
5. Patients with concurrent malignant tumors requiring treatment
6. Patients with active heart disease defined as one or more of the following: (1) Uncontrolled or symptomatic angina pectoris;(2) A myocardial infarction 6 months before enrolled; (3)Arrhythmia needed medication or with severe clinical symptoms;(4)Uncontrolled or symptomatic congestive heart failure (NYHA> grade 2);(5)Left ventricular ejection fraction below the lower limit of the normal range.
7. Uncontrolled active serious infections that could, in the investigator's opinion, potentially interfere with the completion of treatment

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to approximately 2 years
  It is defined as the time from the start of randomization to the occurrence of induction failure or disease progression or death from any cause (whichever occurs first).

SECONDARY OUTCOMES:
Complete remission (CR) rate or complete remission with partial hematologic recovery (CRh) rate or complete remission with incomplete hematologic recovery (CRi) rate | Up to approximately eight weeks
  Proportion of patients with CR, CRh or CRi
Minimal residual disease (MRD)-negative remission rates after induction | Up to approximately eight weeks
  Among those who have achieved CR/CRh/CRi after induction, proportion of patients who is MRD-negative
Cumulative incidence of minimal residual disease (MRD)-negative remission rates | Up to approximately 1 years
  The proportion of patients with negative MRD results at any time during treatment
Relapse-free Survival (RFS) | Up to approximately 2 years
  It is defined as the time from the start of achieving remission to disease progression, death from any cause or the last follow-up.
Overall survival (OS) | Up to approximately 2 years
  It is defined as the time from the start of randomization to the death from any cause.
30-day postinduction mortality | Up to approximately 30 days
  It is defined as death from any cause within 30 days after the start of induction.
60-day postinduction mortality | Up to approximately 60 days
  It is defined as death from any cause within 60 days after the start of induction.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wei, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided